CLINICAL TRIAL: NCT06166017
Title: Lingual Keratinized Tissue in Fully Edentulous Patients and Its Impact on Implant Health
Status: Not yet recruiting | Type: Observational
Sponsor: George Eastman Dental Hospital, Italy (Other)
Responsible Party: Principal Investigator, Lucrezia Paternò Holtzman, Faculty, Senior Researcher, Clinical Professor, George Eastman Dental Hospital, Italy
Other Study IDs: GeorgeEastmanDH
Record Dates: First submitted 2023-11-22; First posted 2023-12-12 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Peri-Implantitis; Peri-implant Mucositis; Recession, Gingival
MeSH Terms: conditions — Peri-Implantitis; Gingival Recession

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Full-arch implant-supported restorations for fully edentulous patients: No interventions will be administered. Instead, clinical parameters will be collected (see detailed description) as well as radiographs of the implants.
  Interventions: Other: Exposure to minimal amount of lingual keratinized tissue width

INTERVENTIONS:
Other: Exposure to minimal amount of lingual keratinized tissue width — measurement of clinical parameters

SUMMARY:
Cross-sectional study involving the measurement of the width of lingual keratinized tissue (in the implant locations) in fully edentulous patients restored with dental implants. The width of KT will be correlated with the primary outcome, diagnosis of peri-implantitis, defined as Probing depth (PPD)>= 6 mm, inflammation/ bleeding on probing (BOP) and bone loss >= 3 mm from the implant platform.

DETAILED DESCRIPTION:
The study will be conducted with a cross-sectional design. All clinical parameters (width of buccal and lingual keratinized tissue, probing depth, bleeding on probing, plaque, crestal bone loss, gingival index, suppuration) will be collected in mandibular implants in fully edentulous lower arches. The width of lingual band of keratinized tissue (KT) will be be correlated with diagnosis of peri-implantitis or peri-implant mucositis.

ELIGIBILITY:
Inclusion Criteria:

* Osseointegrated (non-mobile) and loaded dental implant
* Mandibular implants
* Full-arch implant-supported prostheses
* Removable full-arch prostheses
* Fixed full-arch prostheses

Exclusion Criteria:

* Implants loaded less than 12 months before examination
* Mobile (non integrated) implants
* Partially edentulous patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers presenting with integrated implants supporting a fixed or removable full-arch prosthesis. Minimum loading time of 12 months.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of peri-implantitis (composite outcome made of different outcomes): yes or no (dichotomous) | Day 1
  dichotomous (yes or no) outcome composed by PPD (mm), BoP/SOP (yes or no dichotomous) and bone loss (mm, assessed on radiograph)

SECONDARY OUTCOMES:
Mucosal recession | Day 1
  Distance (mm) between the prosthetic margin/ locator and the mucosal margin
Bleeding on probing (BOP) | Day 1
  dichotomous measure of mucosal inflammation detected via periodontal probe
Probing pocket depth (PPD) | Day 1
  distance between the mucosal margin and the bottom of the sulcus/ pocket (mm)
Self-assessed Brushing discomfort | Day 1
  Rated by patient on Visual analog score (100 mm) to define the amount of discomfort during brushing, with 0 being the minimum and 100 being maximum discomfort. The patient will be asked to rate their level of discomfort by placing an X over the line. The distance from 0 to the X will be measured and converted into a percentage of the entire length of the line.
Crestal bone loss (mm) | Day 1
  Measured on radiograph (in mm) between the implant shoulder and the most coronal location of the crestal bone
Suppuration on probing | Day 1
  measured dichotomously (yes/no) when probing an implant
Diagnosis of mucositis | Day 1
  dichotomous (yes/no) presence of mucosal peri-implant inflammation in the absence of crestal bone loss

IPD SHARING:
Plan to Share IPD: No